CLINICAL TRIAL: NCT00786552
Title: Phase 2 Trial of Pemetrexed (Alimta™) Combined With Paclitaxel in Patients With Recurrent/Advanced Follicular, Papillary or Anaplastic Thyroid Cancer
Brief Title: Pemetrexed + Paclitaxel in Patients With Recurrent/Advanced Thyroid Cancer
Acronym: Panthera
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Prof. Dr. med. J. T. Hartmann, University of Kiel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Panthera
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Thyroid Cancer
Keywords: recurrent/advanced thyroid cancer; papillary or anaplastic thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Recurrence; Thyroid Carcinoma, Anaplastic | interventions — Pemetrexed; Paclitaxel

ARMS (1):
- chemotherapy (Experimental)
  Interventions: Drug: pemetrexed + paclitaxel

INTERVENTIONS:
Drug: pemetrexed + paclitaxel — Pemetrexed 500 mg/m² i.v. over 10 minutes on day 8 Paclitaxel 90 mg/m² i.v. over 60 minutes on day1 and 8

SUMMARY:
The aims of this trial are to evaluate the efficacy and tolerability of pemetrexed + paclitaxel in patients with recurrent/advanced follicular, papillary or anaplastic thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic, histologically proven follicular/papillary or anaplastic thyroid cancer without clinically meaningful surgical or radiotherapeutic options and/or no amenability for radio-iodine therapy and evidence of progressive or symptomatic disease.
* No other forms of chemotherapy or investigational anticancer agents therapy for at least 4 weeks before enrollment in study.
* Performance status of 0 to 2 on the ECOG scale.
* Evidence of measurable disease according to the RECIST criteria.
* Prior radiation therapy and surgery allowed if completed at least 2 weeks prior to study enrollment, prior radioiodine treatment at least 3 months prior to study enrollment and patients must have recovered from the acute toxic effects of the treatment prior to study entry.
* Adequate organ function.
* No active infection (at the discretion of the investigator) or current central nervous system (CNS) metastases or history of central nervous system metastases or other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
* No breast feeding nor pregnancy. For women of childbearing potential a negative serum pregnancy-test has to be performed 7 days prior to inclusion into the study.
* No coexisting second malignancy or history of prior malignancy within the last 5 years. (Excluding basal or squamous cell carcinoma of the skin, superficial bladder cancer and in situ carcinoma of the cervix with no evidence of recurrence).
* For men and women of childbearing potential appropriate contraceptive precautions should be taken during the trial and for 3 months afterwards.
* No significant cardiovascular disease in the form of abnormal electrocardiogram (ECG) coupled with clinical features of recent or recurrent symptomatic cardiac disease (including myocardial infarction within the last year, uncontrolled angina, arrhythmia or hypertension, severe congestive heart failure (NYHA >3)).
* No evidence of peripheral neuropathy greater than CTC Grade 1.
* No prior taxane and/or pemetrexed therapy.
* Ability to discontinue administration of acetysalicylate and other nonsteroidal anti-inflammatory agents (NSAID) for 2 days before, the day of, and 2 days after the dose of pemetrexed (5 days prior for long-acting agents such as piroxicam). Exceptions for selective cyclooxygenase II-inhibitors in analgesic treatment may be discussed.
* No clinically significant effusions (pleural or peritoneal), or albumin <2.5 g/dl at the time of study treatment application. The drainage of effusions prior to study treatment application is possible.
* Inability of oral intake of folic acid or intramuscular vitamin B12 supplementation.
* At least 18 years of age and absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.
* Participation in another trial at the same time is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Rate of response | 6 weeks

SECONDARY OUTCOMES:
Toxicity | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Joerg T Hartmann, MD, Principal Investigator — Medical Center II, University of Kiel, Germany
Locations (1):
- Medical Center II, University of Kiel, Kiel, Germany